CLINICAL TRIAL: NCT06934460
Title: A Randomised Clinical Study on Indirect Lithium Disilicate Versus Direct Composite Restorations in Severely Compromised Endodontically Treated Molar Teeth
Brief Title: Direct Versus Indirect Endocrowns on Endodontically Treated Molars
Acronym: Endocrowns
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201500425
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Endodontically-Treated Teeth; Endocrown Restoration; Restoration of Posterior Teeth; Composite Resins
Keywords: endocrown; endocrown restoration; composite resin; direct composite; endodontically-treated teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial comparing direct composite resin and lithium disilicate endocrowns on endodontically treated molar teeth.
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct composite resin endocrown (Active Comparator): Direct restoration with a microhybrid composite resin
  Interventions: Device: Composite resin
- Lithium disilicate endocrown (Experimental): Indirect restoration with a lithium disilicate endocrown in conjunction with Immediate Dentin Sealing
  Interventions: Device: lithium disilicate endocrown

INTERVENTIONS:
Device: Composite resin — Direct composite resin restoration after application of an adhesive system
  Arms: Direct composite resin endocrown
Device: lithium disilicate endocrown — Lithium disilicate endocrown in conjunction with Immediate Dentin Sealing
  Arms: Lithium disilicate endocrown

SUMMARY:
In this clinical trial the performance of monolithic restorations made of indirect lithium disilicate ceramic and direct resin composite materials on severe structurally compromised endodontically treated molar teeth is evaluated.

Rationale: It is presumed that indirect restoration of extensively restored endodontically treated molar teeth contributes to durability. However, there is a lack of evidence concerning the performance of both indirect ceramic and direct composite monolithic restorations. Such restorations are commonly named 'endocrowns'.

Objective: The objective of the study is to investigate which treatment modality, indirect ceramic or direct composite endocrowns, provide the best restoration of severe structurally compromised endodontically treated molar teeth in terms of clinical performance.

Study design: Randomised 5-year clinical trial with endodontically treated molar teeth restored with either indirect glass ceramic (experimental) or direct resin composite endocrowns (control).

Study population: A total of 102 severe structurally compromised endodontically treated molar teeth that need to be restored, with a maximum of two restorations per patiënt. Patients are healthy volunteers over 18 years.

Intervention: Each patiënt with a restorative indication for endodontically treated first and second molar teeth will be randomly assigned to one of two treatment groups: indirect glass ceramic endocrown or direct composite endocrown.

DETAILED DESCRIPTION:
In this clinical trial the performance of monolithic restorations made of indirect lithium disilicate ceramic and direct resin composite materials on severe structurally compromised endodontically treated molar teeth is evaluated.

Rationale: It is presumed that indirect restoration of extensively restored endodontically treated molar teeth contributes to durability. However, there is a lack of evidence concerning the performance of both indirect ceramic and direct composite monolithic restorations. Such restorations are commonly named 'endocrowns'.

Objective: The objective of the study is to investigate which treatment modality, indirect ceramic or direct composite endocrowns, provide the best restoration of severe structurally compromised endodontically treated molar teeth in terms of clinical performance.

Study design: Randomised 5-year clinical trial with endodontically treated molar teeth restored with either indirect glass ceramic (experimental) or direct resin composite endocrowns (control).

Study population: A total of 102 severe structurally compromised endodontically treated molar teeth that need to be restored, with a maximum of two restorations per patiënt. Patients are healthy volunteers over 18 years.

Intervention: Each patiënt with a restorative indication for endodontically treated first and second molar teeth will be randomly assigned to one of two treatment groups: indirect glass ceramic endocrown or direct composite endocrown.

ELIGIBILITY:
Inclusion Criteria:

ASA i or II [de Jong, 1994], This ASA score is already known before participation, due to regular check-ups.

* Asymptomatic endodontically treated and heavily restored upper and lower molar teeth with an indication for a (new) restoration.
* Pulp chamber height of at least 2 millimeters.
* Need of cuspal coverage;
* Pockets around the molar 3-5 mm.
* Moderate to low caries risk.

Exclusion Criteria:

* ASA III or higher.

  * Pockets around the molar >5mm.
  * Presence of an accessible furcation.
  * No biological width present (3mm).
  * Rubber dam placement not possible.
  * No antagonistic tooth.
  * History of severe parafunction.
  * High caries risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Restoration survival | 5 years
  Failure is defined as restoration replacement or tooth extraction due to secondary decay or vertical root fracture (FDI scre 5). A FDI score of 4 or less indicates survival.

SECONDARY OUTCOMES:
Abutment tooth survival | 5 years
  Failure defined as tooth extraction, regardless of cause.

OTHER OUTCOMES:
Abutment tooth success | 5 years
  failure was defined as tooth extraction, the presence of endodontic pathology, or the necessity for (non-)surgical endodontic retreatment
Patient satisfaction | 1 and 5 years
  Patient satisfaction measured on VAS-scale (0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Marco S. Cune, Prof.dr., Study Director — Department of Restorative Dentistry and Biomaterials - Center for Dentistry and Oral Hygiene - University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: Undecided
Start before 2019 with the inclusion and was not mentioned in informed consent forms specifically